CLINICAL TRIAL: NCT07050498
Title: Evaluation of the Effects of Virtual Reality on Preoperative Anxiety in Refractive Surgery
Acronym: ERVAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A01771-44
Record Dates: First submitted 2025-06-04; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Refractive Disorders
Keywords: refractive surgery
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, randomized, open-label study on two parallel groups of patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): Preoperative conditioning by virtual reality + Routine preoperative procedure (local anesthesia)
  Interventions: Device: Virtual reality
- Usual care (Active Comparator): Routine preoperative procedure (local anesthesia)
  Interventions: Procedure: Usual Care Group

INTERVENTIONS:
Device: Virtual reality — Virtual reality hypnosis software applications are Class I medical devices according to Rule 12 of Directive 93/42/EC. They allow, through a virtual reality headset and headphones, to immerse the patient in a hypnotic sound and visual environment. Several visual scenarios can be proposed, allowing the patient to virtually travel to a beach, the seabed, on an alpine walk, etc.).
  The HypnoVR Biofeedback virtual reality device is provided by the HypnoVR company.
  Arms: Virtual reality
Procedure: Usual Care Group — Routine preoperative procedure (local anesthesia)
  Arms: Usual care

SUMMARY:
The objective of this study is to determine to what extent the use of a software application prior to refractive surgery involving multisensory immersion (visual and auditory) in a hypnotic and relaxing sound and visual environment can reduce anxiety levels.

The assessment of preoperative anxiety levels will be based on the administration of a psychometric scale (APAIS scale) and the measurement of salivary cortisol, which is a sensitive marker of the patient's stress level.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, single-center study conducted on two parallel groups of patients undergoing refractive surgery (virtual reality preoperative conditioning or routine preoperative procedure). Therapeutic benefit is based on the assessment of preoperative anxiety using the APAIS scale.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older,
* Patient who has read and signed the consent form for participation in the study after a reflection period (between 10 and 45 minutes)
* Patient who is a candidate for refractive surgery

Exclusion Criteria:

* Contraindication to virtual reality (uncontrolled epilepsy, hearing impairment)
* Pregnant or breastfeeding patient
* Cushing's disease, Addison's disease, hypo- or hyperthyroidism
* Patient treated with topical or systemic corticosteroids
* Patient treated with neuroleptics, anxiolytics, or antidepressants
* Patient under legal protection, guardianship, or curatorship
* Patient participating in another blinded research study
* Patient not affiliated with the French social security system
* Patient unable to understand the information provided and/or give written informed consent: dementia, psychosis, impaired consciousness, non-French-speaking patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Preoperative anxiety level | Preoperative procedure
  The preoperative anxiety level is measured on the APAIS scale. The APAIS scale is a self-assessment consisting of six questions with expected responses rated from 1 (the patient strongly disagrees with the statement) to 5 (the patient strongly agrees with the statement) out of a minimum overall score of 6 and a maximum overall score of 30. The first three questions relate to anesthesia, and the next three relate to surgery. Of the three questions (related to anesthesia or surgery), two assess preoperative anxiety, and the third assesses the need for information.
  The APAIS scale calculates four scores: overall anxiety, surgery-related anxiety, anesthesia-related anxiety, and information need. A total anxiety score of 11 or higher corresponds to a high level of anxiety.

SECONDARY OUTCOMES:
Intraoperative pain intensity | Immediately after surgery
  Pain intensity will be assessed using a simple numerical rating scale (SNR) ranging from 0 (no pain) to 10 (worst imaginable pain).
Postoperative pain intensity | 15 minutes after the End of surgery
  Pain intensity will be assessed using a simple numerical rating scale (SNR) ranging from 0 (no pain) to 10 (worst imaginable pain).
Intraoperative comfort | 15 minutes after the End surgery
  Comfort will be assessed using a simple numerical rating scale (SNR) ranging from 0 (minimum comfort) to 10 (maximum comfort).
Postoperative Overall Patient Satisfaction | 15 minutes after the End of surgery
  Overall Patient Satisfaction will be assessed using a simple numerical rating scale (SNR) ranging from 0 (not at all satisfied) to 10 (very satisfied).
Change in salivary cortisol | Before any study procedure
  After rinsing the mouth with water, a 1 ml sample of salivary secretions without stimulation will be taken using a Salivette® (Sarstedt TM). The samples will be stored at -20°C before being analyzed by the private laboratory Eurofins, using an ELISA test (analytical sensitivity = 1.38 nmol/L; functional sensitivity = 8.28 nmol/L; upper detection limit ~110 nmol/L).
Change in salivary cortisol | Just before surgery
  After rinsing the mouth with water, a 1 ml sample of salivary secretions without stimulation will be taken using a Salivette® (Sarstedt TM). The samples will be stored at -20°C before being analyzed by the private laboratory Eurofins, using an ELISA test (analytical sensitivity = 1.38 nmol/L; functional sensitivity = 8.28 nmol/L; upper detection limit ~110 nmol/L).
Change in salivary cortisol | 15 minutes after the end of surgery
  After rinsing the mouth with water, a 1 ml sample of salivary secretions without stimulation will be taken using a Salivette® (Sarstedt TM). The samples will be stored at -20°C before being analyzed by the private laboratory Eurofins, using an ELISA test (analytical sensitivity = 1.38 nmol/L; functional sensitivity = 8.28 nmol/L; upper detection limit ~110 nmol/L).
Heart rate | Before any study procedure
  Heart rate measurement in both groups
Blood pressure | Before any study procedure
  Blood pressure measurement in both groups
Heart rate | Before surgery
  Heart rate measurement in both groups
Blood pressure | Before surgery
  Blood pressure measurement in both groups
Heart rate | 15 minutes after the end of surgery
  Heart rate measurement in both groups
Blood pressure | 15 minutes after the end of surgery
  Blood pressure measurement in both groups
Tolerance | 15 minutes after the end of surgery
  The tolerance of the test procedure will be assessed by collecting adverse events occurring during the duration of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Monticelli, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided